CLINICAL TRIAL: NCT00933296
Title: Schnitzler Syndrome: Clinical Study, Physiopathological and Search for Genetic
Brief Title: Schnitzler Syndrome: Clinical Study, Physiopathological and Search for Genetic Factors
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 4350
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Schnitzler Syndrome
Keywords: Schnitzler syndrome; Waldentsröm's disease; anakinra
MeSH Terms: conditions — Schnitzler Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — White cells Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A Patients with the Schnitzler syndrome: Patients with the Schnitzler syndrome
- B Control subjects:: B1 healthy B2 other diseases

SUMMARY:
The Schnitzler syndrome is a rare entity characterized by an urticarial rash and recurrent fever in a patient with a monoclonal IgM component. Other frequent signs include joint, bone and muscle pain, enlarged spleen, liver and lymph nodes, increased blood sedimentation rate (BSR), elevated neutrophil count and abnormalities on bone morphologic investigations. In 2001, the investigators proposed criteria to diagnose this syndrome, which are currently admitted in the literature. The main complications of the Schnitzler syndrome are a difficult-to-control inflammatory anemia, AA-amyloidosis and malignant B lymphoproliferative disorders. About 15% of patients with a Schnitzler will eventually develop a lymphoproliferative disorder; thus this syndrome allows studying the relationship between lymphomagenesis and inflammation. By many aspects, the Schnitzler syndrome is reminiscent of auto-inflammatory syndromes. Though the term auto-inflammatory disease is as to yet restricted to diseases with Mendelian inheritance, some polygenic inflammatory diseases like for example Crohn's disease clearly involve pathogenetic pathways shared with the monogenic auto-inflammatory syndromes. The investigators stipulate that this could also be the case in the Schnitzler syndrome for the following reasons: (1) this is a recurrent fever of unknown cause; (2) the peculiar eruption, characterized pathologically by a neutrophilic infiltrate very similar to the one observed in the auto-inflammatory cryopyrinopathies (CINCA/NOMID syndrome, Muckle-Wells syndrome and familial cold-urticaria); the investigators recently individualized this particular eruption, significantly associated with systemic inflammatory disease, within the group of neutrophilic urticarias (Kieffer et al. Medicine, in press); (3) the occurrence of aseptic neutrophilic osteitis, very similar to the one reported in patients with Majeed syndrome, another auto-inflammatory syndrome; (4) a significant increase of neutrophil count, not otherwise explained; (5) a spectacular response to the IL-1 inhibitor, within hours after the first injection, similar to what is reported in the PAPA (pyogenic arthritis, pyoderma gangrenosum and acne) syndrome or the cryopyrinopathies, suggesting a direct pathogenic effect of IL-1.

ELIGIBILITY:
Inclusion Criteria:

* patients with the Schnitzler syndrome according to criteria established by Lipsker D et al. Medicine (Baltimore) 2001;80:37-44

Exclusion Criteria:

* children and pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: University hospitals
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2009-07; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Lipsker, Pr, Principal Investigator — HUS
Locations (17):
- France (15):
  - CHU de Besançon Service de Dermatologie, Besançon
  - Service de DermatologieCHU Morvan5 avenue Foch, Brest
  - Centre Hospitalier Général Bd Yves du Manoir, Dax
  - Service de Rhumatologie Centre Hospitalier du Mans, Le Mans
  - Service de Médecine Interne Hôpital Claude-Huriez, Lille
  - Service de DermatologieHôtel Dieu, Lyon
  - Service médecine interne et thérapeutique Hôpital sainte marguerite, Marseille
  - Service de Dermatologie Hôpital Saint Eloi 80 avenue A Fliche, Montpellier
  - Service de dermatologie CHU Hôtel Dieu1 place Alexis Ricordeau, Nantes
  - Unité de médecine interne Centre Hospitalier G. Renon, Niort
  - Service d'immuno-hématologie Hôpital St-Louis 1 av Claude Vellefaux, Paris
  - Service de médecine interne Hôpital Tenon4, rue de la Chine, Paris
  - Service de dermatologieCHU GUERIN2 rue de la Milétrie, Poitiers
  - BOYE Thierry, Toulon
  - Service de médecine interne-néphrologie Centre Hospitalier Valenciennes, Valenciennes
- Italy (2):
  - Azienda Ospedaliero Universitaria Policlinico, Bari
  - Clinica DermatologicaUnivesité de GênesVialle Benedetto, Genova